CLINICAL TRIAL: NCT05140629
Title: Adansonia Digitata L. (Baobab Fruit) Effect on Postprandial Glycaemia in Healthy Adults: a Randomized Controlled Trial
Brief Title: Effect of Baobab Fruit on Postprandial Glycaemia in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 518baobab
Record Dates: First submitted 2021-11-05; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Hyperglycemia, Postprandial
Keywords: Adansonia digitata; Baobab fruit; Postprandial glycaemia; Antioxidant; Polyphenols; Proanthocyanidins
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (OGTT) (Placebo Comparator): The control group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the ADA, dissolved in 200 ml of water.
  Interventions: Other: Placebo OGTT
- Intervention (OGTT plus Baobab fruit extract) (Experimental): The intervention group ingested glucose solution followed by 250 ml of baobab aqueous extract (33.33 g FW).
  Interventions: Other: Baobab fruit aqueous extract

INTERVENTIONS:
Other: Baobab fruit aqueous extract — After overnight fasting, blood glucose level was assessed through a capillary drop blood, immediately before Oral Glucose Tolerance Test (t0). The intervention group ingested glucose solution followed by 250 ml of baobab aqueous extract (33.33 g FW). Blood glucose level was also measured at 30 (t30), 60 (t60), 90 (t90) and 120 (t120) minutes immediately after intervention, for each participant, in control and intervention groups. Glucometer equipment, strips for glucose meters (One Touch Select Plus) and sterilized lancets (Sarstedt normal 21G) were used to measure blood glucose concentrations, taking due care of safety and asepsis.
  Arms: Intervention (OGTT plus Baobab fruit extract)
Other: Placebo OGTT — After overnight fasting, blood glucose level was assessed through a capillary drop blood, immediately before Oral Glucose Tolerance Test (t0). The control group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the ADA, dissolved in 200 ml of water. Blood glucose level was also measured at 30 (t30), 60 (t60), 90 (t90) and 120 (t120) minutes immediately after intervention, for each participant, in control and intervention groups. Glucometer equipment, strips for glucose meters (One Touch Select Plus) and sterilized lancets (Sarstedt normal 21G) were used to measure blood glucose concentrations, taking due care of safety and asepsis.
  Arms: Placebo (OGTT)

SUMMARY:
Baobab fruits have been traditionally used in Africa due to its therapeutic proprieties attributed to it high polyphenol content. The aim of the study was to investigate the effect of baobab fruit on postprandial glycaemia on healthy adults and to measure its bioactive compounds and antioxidant activity. The study was conducted on 31 healthy subjects. The participants were randomly allocated in control group (oral glucose tolerance test (OGTT); n = 16) and in intervention group (OGTT followed by administration of 250 ml baobab aqueous extract (BAE); n = 15). Total phenols, proanthocyanidins, hydrolysable tannins and antioxidant activity (FRAP, DPPH, ABTS and inhibition of O2•- and NO• methods) were quantified. Repeated Measures ANOVA of mixed type and Independent samples t-test were used.

DETAILED DESCRIPTION:
This study was approved by Egas Moniz Cooperativa de Ensino Superior Ethics Committee (protocol code 518) and was carried out in accordance with the Declaration of Helsinki (Declaration of 1975, revised in 2000). An informed consent was given to all eligible participants, after oral and written information about the study.

This randomized controlled clinical trial, blind to subjects, was conducted with 31 subjects, recruited at the Campus Universitário Egas Moniz, in Monte de Caparica, Portugal. After eligibility criteria and inform consent signed, participants were subjected to the inclusion and exclusion criteria and subsequently randomly allocated in to control or intervention groups. The method of allocation sequence was based on sequentially numbers. The first patient was randomly assigned to intervention or control group, and the following patients were sequentially allocated alternately to each group. A codification was attributed to each participant in order to maintained anonymity and ensure confidentiality of data.

After a period of 8-10 hours fasting, the control group was given OGTT and the intervention group was given OGTT followed by baobab aqueous extract.

Baobab aqueous extract preparation:

The baobab fruit was bought in the market of Benfica, located in the city of Luanda (Angola) and brought to Lisbon (Portugal) duly packed in a plastic bag and stored in a dried environmental local until needed. For the aqueous extraction of the fruit 40 ± 1 g of pulp, seeds and red filaments were weighed and the fruit was boiled in 300 ml of water for 5 minutes. After slowly cooling until room temperature, extract was then placed in a refrigerator in a container where it remained for 8 hours at an average temperature of 10°C. The BAE was sieved with the aid of a net sieve, separating it from the seeds and filaments, and was subsequently subjected to the clinical trial and the antioxidant assays. For the antioxidant assays, after filtration, the extract was passed through the blender (Kenwood Multipro Compact Food Processor FDP302SI), filtered again obtaining homogeneous samples, avoiding the formation of precipitates during the analysis. Final concentration of the aqueous extract obtained, for both clinical trial and chemical analysis, was 0.1333 g Adansonia digitata L. (AD) / ml extract fresh weight (FW).

Interventions:

After overnight fasting, blood glucose level was assessed through a capillary drop blood, immediately before Oral Glucose Tolerance Test (t0). The control group participants ingested glucose solution alone (OGTT) prepared with 75 g of anhydrous oral glucose as prescribed by the American Dietetic Association (ADA), dissolved in 200 ml of water. The intervention group ingested glucose solution followed by 250 ml of baobab aqueous extract (33.33 g FW). Blood glucose level was also measured at 30 (t30), 60 (t60), 90 (t90) and 120 (t120) minutes immediately after intervention, for each participant, in control and intervention groups. Glucometer equipment, strips for glucose meters (One Touch Select Plus) and sterilized lancets (Sarstedt normal 21G) were used to measure blood glucose concentrations, taking due care of safety and asepsis. Based on the glycaemia values, the blood glucose incremental area under the curve (AUCi) of each participant was defined using the GraphPad Prism program (version 5.0). Maximum concentrations (Cmax) and variations of maximum concentrations (ΔCmax) were determined by comparing them with their respective baseline glycemia levels values.

Anthropometric parameters assessment:

The anthropometric parameters were also collected, namely, weight, height and body mass index (BMI). The BMI was calculated as weight (Kg) divided by height (m2) squared (Kg/m2). Body weight was estimated by bio-impedance, through scale the Inbody®, model 230.

Dietary ingestion assessment:

Participants of the study completed a 24-hour food recall questionnaire, which were carefully instructed by an investigator to identify all food consumed. The amount of each food ingested was estimated with help from pictures. A book with pictures of meals in different sizes was used. The investigator reviewed the questionnaire together with the participant. Food intake of each participant was analysed using the software The Food Processor SQL (version 11.3.285) obtaining total energy, carbohydrates, proteins and lipids mean intake.

Total phenol, proanthocyanidins and hydrolysable tannins content assessment:

Total phenolic concentration was determined according to the Folin Ciocalteu method employing gallic acid as standard. Results were expressed as mg of gallic acid equivalents/L (GAE/L). For this analysis, 125 μl of BAE, previously diluted (x15) in water and 125 μl of ethanol was added to 2.5 ml of Folin-Ciocalteu reagent solution (1:10 diluted in H2O) and 2 ml of aqueous sodium carbonate (Na2CO3) 1M. After 15 minutes the absorbance was measured at 765 nm.

The content of proanthocyanidins was determined according to Gu et al (2002) method with modifications, which is based on acidic hydrolysis of proanthocyanidins polymers producing reddish pigments in hot 1-butanol/ hydrochloric acid solution. It was added 200 μl of BAE diluted (x2) to 200 μl of methanol and 2600 μl of HCl /1-butanol 10%(v/v) solution. The test tubes were shaken and incubated, at 100°C for 50 minutes. The absorbance was measured at 550 nm. Results are expressed as mg equivalents of proanthocyanidins A2 /L (EPA2/L).

The method of Willis and Allen was adapted for the determination of hydrolysable tannins of the BAE. A volume of 1 ml of extract was added to 5 ml of 2.5% potassium iodate (KIO3). The mixture was then stirred and returned to the water bath at 25°C for 20 minutes. Absorbance reading was performed by a spectrophotometer at 550 nm and the results were expressed as mg of tannic acid equivalents/L (TAE/L).

Antioxidant assays:

Ferric Reducing Antioxidant Power (FRAP) method: the antioxidant effect (reducing ability) was evaluated by monitoring the formation of an intense blue color from the Fe2+ TPTZ complex, according to the Ferric Reducing Antioxidant Power (FRAP) assay. A volume of 2850µl (25ml 300mM acetate buffer pH=3,6 solution plus 2,5 ml 10mM TPTZ solution in HCl 40mM + 2,5 ml 20mM FeCl3.6H2O solution) was added to 150µl of diluted BAE.. The tubes were kept in the dark for 30 minutes (7 assays at different concentrations). The absorbance was determined at 593 nm and the results were expressed in mg of Trolox equivalents/L (TE/L).

ABTS method: this method was based on the capacity of a sample to inhibit the ABTS radical (ABTS+) compared with a reference antioxidant standard (Trolox). The ABTS+ radical was generated by chemical reaction with potassium persulfate (K2S2O8). Thus, 25 ml of ABTS (7 mM) was added to 440 µl of K2S2O8 (140 mM) and allowed to stand in darkness at room temperature for 12-16 h. The solution was prepared by taking a volume of the previous solution and diluting it in ethanol until its absorbance at λ = 734 nm was 0.70. The tubes were kept in the dark for 30 minutes. The results expressed in mg of Trolox equivalents/L (TE/L).

The DPPH method: this method was determined by the 2,2-diphenyl-1-picrylhydrazyl radical scavenger. A volume of 150 μl BAE was added to 2850 μl of DPPH solution previously prepared in methanol with a λ=515 nm of 1.1. The solutions were kept for 24 hours in the absence of light. The absorbance was determined at 515 nm and the results expressed in mg of Trolox equivalents/L (TE/L).

Inhibition capacity of O2•- anion and NO radical:

The superoxide anion is generated by oxidation of NADH by reacting with PMS and oxygen, causing the reduction of NBT. A volume of 500 μl of BAE with different concentration were added to 2 ml of NADH (189μM) and NBT (120 μM) in 40 mM Tris-HCl buffer pH 8. The reaction was started after the addition of 0.5 ml of PMS (60 μM) and after 5 minutes incubation at room temperature, the absorbance was measured at 560 nm.

The inhibition NO radical test was based on the method of Nikkhah and coworkers (2008). A volume of 250 μl of BAE with different concentrations was added to 1 ml of sodium nitroprusside and 250 μl of phosphate buffered saline (PBS). The mixture was kept for 150 minutes at 25°C. Then, 0.5 ml of this mixture was added to 1 ml of sulfanilic acid (0.33% in 20% glacial acetic acid), and kept for 5 minutes at room temperature. Then it was added 1 ml of NED (0.1% w/v) and kept this mixture for 30 minutes at 25°C. At the end of the reaction a pink chromophore was formed. The absorbance was measured at 540 nm. The percentage of inhibition of O2•- and NO radicals was determined using equation 1 and the results were expressed as mg of gallic acid equivalents (GAE)/L.

Statistical analysis:

Statistical analysis was performed using the Excel® and SPSS® (Statistical Package for Social Sciences) version 27.0 software for Mac. Data are presented as mean ± SD (standard deviation) and SEM (standard error of the mean). Repeated measurement ANOVA of mixed type was used to assess the difference between the 2 groups for postprandial blood glucose at different times. The independent samples t-test was used to assess the difference between the 2 groups for anthropometric parameters, total energy intake, carbohydrates, protein and lipid, Cmax, ΔCmax and AUCi values. All statistical tests were performed at the 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Not currently undergoing lactation or pregnancy,
* To be able to read and sign the informed consent.
* Healthy subjects and a fasting blood glucose < 126 mg/dl

Exclusion Criteria:

* Subjects that were less than 8 or more than 10 hours fasting,
* To have symptoms and history of gastrointestinal, hepatic and cardiovascular diseases
* Baobab intolerance or allergy,
* Drug and/or supplement consumption capable of influencing plasma glucose
* Have ingested baobab, water, coffee or alcohol intake and smoked tobacco consumption within 8 hours before the intervention

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose levels time curve | Before intervention and after 30, 60, 90, and 120 minutes after intervention
  Mean blood glucose levels (mmol/L) obtained after oral glucose tolerance test in control group and after oral glucose tolerance test plus baobab extract in intervention group at different moments
Incremental area under the curve of glucose levels | At 120 minutes after intervention
  the blood glucose incremental area under the curve (AUCi) of each participant was defined using the GraphPad Prism program (version 5.0).
Blood glucose maximum concentrations | At 120 minutes after intervention
  Mean blood glucose levels (mmol/L)

SECONDARY OUTCOMES:
Weight of participants | At baseline
  Mean values of weight (in kilograms)
Body mass index of participants | At baseline
  Mean values of body mass index (Kg/m2), calculated as weight (Kg) divided by height (m2) squared (Kg/m2)
Height of participants | At baseline
  Mean values of height (in meters)
Total energy intake intake of participants | At the day before intervention
  Mean values of total energy intake (in kilocalorie - Kcal), obtained through The Food Processor SQL software
Total protein intake of participants | At the day before intervention
  Total protein intake (in grams - g), obtained through The Food Processor SQL software
Total carbohydrate intake of participants | At the day before intervention
  Total carbohydrate intake (in grams - g), obtained through The Food Processor SQL software
Total lipid intake of participants | At the day before intervention
  Total lipid intake (in grams - g), obtained through The Food Processor SQL software
Total phenols content determination | At baseline
  Mean values of total phenols (expressed as mg of gallic acid equivalents/L - GAE/L)
Proanthocyanidins content determination | At baseline
  Mean values of proanthocyanidins (expressed as mg equivalents of procyanidin A2 /L - EPA2/L)
Hydrolysable tannins content determination | At baseline
  Mean values of hydrolysable tannins (expressed as mg of tannic acid equivalents/L - TAE/L)
DPPH radical scavenger capacity | At baseline
  Mean values of antioxidant capacity by DPPH (2,2-diphenyl-1-picrylhydrazyl) radical scavenger (expressed in mg of Trolox equivalents/L - TE/L)
Ferric Reducing Antioxidant Power (FRAP) determination | At baseline
  Mean values of antioxidant capacity by FRAP test (expressed in mg of Trolox equivalents/L - TE/L).
ABTS radical (ABTS+) inhibition capacity | At baseline
  Mean values of ABTS inhibition capacity (expressed in mg of Trolox equivalents/L - TE/L).
Superoxide radical inhibition capacity | At baseline
  Percentage of superoxide radical inhibition capacity (expressed as %)
Nitric oxide inhibition capacity | At baseline
  Percentage of nitric oxide radical inhibition capacity (expressed as %)

CONTACTS AND LOCATIONS:
Overall Officials: Margarida Moncada, PhD, Principal Investigator — Centro de Investigação Interdisciplinar Egas Moniz, Instituto Universitário Egas Moniz, Portugal
Locations (1):
- Instituto Universitário Egas Moniz, Almada, Monte de Caparica, Portugal